CLINICAL TRIAL: NCT04593355
Title: HCV Epidemiological Survey of Chinese in Northeast Rural Area Which Have Injection History
Brief Title: HCV Epidemiological Survey in China Rural Area
Acronym: HCVES
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Junqi Niu, Vice-President of First Hospital of Jilin University, The First Hospital of Jilin University
Other Study IDs: 20110101
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis
Keywords: Predict; Hepatitis C Virus; Metabolomics
MeSH Terms: conditions — Hepatitis; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood serum,Peripheral blood mononuclear cells (PBMC),Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCV

SUMMARY:
The purpose of this study is to determine whether the morbidity of hepatitis C with Chinese population.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection rate in China is about 3%, which means about 30 million patients. More importantly, many of those patients with chronic hepatitis C eventually develop cirrhosis and hepatocellular carcinoma(HCC).Our survey found the rate of hepatitis c infection in northeastern China without intervention is 34.3%, due to the abuse of caffeine sodium benzoate. This population has the similar mode of transmission, which is a fine study of the natural outcome hepatitis C. We plan to carry out epidemiological studies for this population, review of the influencing factors of the disease, and analyze the host factors that can effect the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* aged from 20 to 65

Exclusion Criteria:

* Has history of decompensated liver diseases
* Has been treated with other anti-virus drugs,or anti-tumor drugs,immuno-suppression drugs
* Has a history of autoimmune hepatitis
* History of a severe seizure disorder or current anticonvulsant use
* History or other evidence of a medical condition associated with chronic liver disease other than HCV which would make the patient, in the opinion of the investigator, unsuitable for the study (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are from the northeast of China. Most of the patients have been infected by the hepatitis c virus due to the drug abuse. Many of them share the same syringe for drug intravenous injection. However, HIV infection has been rarely detected.
Sampling Method: Probability Sample
Enrollment: 6068 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Blood Anti-HCV | Baseline
  Co-infection status are analyzed.

SECONDARY OUTCOMES:
Alanine Aminotransferase (ALT) and Aspartate transaminase (AST) | Baseline
  ALT AST are assayed to detect the hepatic function.
Fibrosis stage | Baseline
  Fibrosis is analyzed with Fibroscan.
Regular blood test | Baseline
  The distribution and absolute count of the different types of blood cells are assayed.
Blood HCV RNA Copies | Baseline
  Blood HCV RNA copies were assayed with Roche - COBAS® AmpliPrep/COBAS® TaqMan® HCV Test.
HCV genotype | Baseline
  HCV NS5A is cloned into T vector and sequenced for evolutionary analysis.
Drug abuse history | Baseline
  Patients will be asked about their drug usage history.
Alcohol ,smoking condition | Baseline
  Patients are asked whether they take alcohol or smoke cigarettes during the therapy period.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, PhD/MD, Study Chair — The First Hospital of Jilin University
Locations (1):
- First Hospital Jilin University, Changchun, Jilin, China